CLINICAL TRIAL: NCT05794295
Title: Sleep Architecture & Cognition in Focal Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2072010
Record Dates: First submitted 2023-02-28; First posted 2023-04-03 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Focal Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Acoustic Stimulation

STUDY DESIGN:
Intervention Model Description: The study is a parallel design with FE patients and healthy controls.
Who Masked: Participant
Masking Description: Participants will not be aware of whether they have acoustic stimulation or sham stimulation. They will be asleep while they are monitored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acoustic Stimulation (AS) (Active Comparator): Participants in this arm will be exposed to acoustic stimulation while they sleep during a night of monitoring.
  Interventions: Other: Acoustic Stimulation (AS)
- SHAM Stimulation (Sham Comparator): Participants in this arm will not be exposed to any stimulation while they have their sleep monitored for one night.
  Interventions: Other: SHAM Stimulation

INTERVENTIONS:
Other: Acoustic Stimulation (AS) — Acoustic Stimulation will be administered while participants have their sleep monitored.
  Arms: Acoustic Stimulation (AS)
Other: SHAM Stimulation — No stimulation will be administered while participants have their sleep monitored.
  Arms: SHAM Stimulation

SUMMARY:
Focal Epilepsy (FE) patients and healthy controls will wear an actigraph at home for one week and a home sleep study device at home for one night. Participants will then undergo two nights of testing (at least one week apart) at California Sleep Solutions (CSS) in Sacramento, CA. During the overnight stays, participants will have EEG leads placed and possibly a headband. They will undergo cognitive testing before they go to sleep and again in the morning. During one night of testing, sounds will be played in the room (acoustic stimulation). The sounds should not wake the participants.

DETAILED DESCRIPTION:
This study will investigate the interconnections between sleep physiology and cognitive deficits in FE and will provide essential pilot data for an interventional trial to characterize the comprehensive effects of AS/ES on sleep and cognition in FE. The long-term goal of this project is to leverage the connections between sleep, behavior, and neural network activity to develop and implement tailored cognitive and sleep interventions for individuals with epilepsy.

AIM 1: Characterize sleep architecture patterns in Focal Epilepsy (FE) and determine the relationship to cognitive processing.

AIM 2: Determine the effect of Sleep Stimulation (Acoustic and/or electrical - AS/ES) on sleep architecture patterns and cognitive processing in FE.

Aim 1 Hypothesis: Compared to controls, FE patients will exhibit interictal epileptiform discharges (IEDs) as well as reduced sleep spindle density and slow wave power with reduced slow wave sleep spindle oscillations (SW-SSO) coupling.

Aim 1 Hypothesis: Compared to controls, reduced SW-SSO coupling during sleep in FE patients will be associated with poorer memory and attention.

Aim 2 Hypothesis: AS/ES will exhibit greater levels of SW-SSO coupling compared to Sham Stimulation.

Aim 2 Hypothesis: Compared to Sham, AS will show increased connectivity on EEG, and improved memory and attention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years of age
* Focal Epilepsy
* Capacity to fully cooperate and follow directions
* no other significant neurological disorders which could affect cognition

Exclusion Criteria:

* Current use of any medications that can significantly affect cognition
* No severe sleep apnea

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Stanford Sleepiness Scale | participant completes over one week post EMU stay
  Alertness Test; charts how alert a participant feels for up to 18 hours of the day for 7 days; scale is from 1-7 with higher scores meaning more sleepiness; abnormal is 4 and above
Pittsburgh Sleep Quality Index (PSQI) | screening
  used to measure quality and patterns of sleep in adults
Epworth Sleepiness Scale | screening
  subjective measure of a patient's sleepiness; scores are from 0-24 with higher scores meaning more sleepiness; abnormal is 10 and above
Karolinska Sleepiness Scale / Sleep Diary | screening
  Self-administered indication of sleepiness; scores are from 1-9 with higher scores meaning more sleepiness; abnormal is 7 and above
Vigor Affect Visual Analog Scale | screening
  self-administered assessment of mood; scores are from 0-10; depending on the question, higher score can mean more sleepiness or less sleepiness

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No